CLINICAL TRIAL: NCT02228850
Title: A Phase 2a Double-Blind, Randomized, Placebo-Controlled Crossover Trial of the Acute Peripheral Vascular Effects, Safety and Tolerability of Alprostadil Topical Cream in Subjects With Raynaud's Phenomenon Secondary to Systemic Sclerosis (SSc, Scleroderma)
Brief Title: Study of Acute Peripheral Vascular Effects, Safety and Tolerability in Subjects With Raynaud's Phenomenon Secondary to Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NexMed (U.S.A.), Inc. (subsidiary of Apricus Biosciences, Inc.) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NexMed 2014-RPS-001
Record Dates: First submitted 2014-08-20; First posted 2014-08-29 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Raynaud's Phenomenon Secondary to Systemic Sclerosis
Keywords: Secondary Raynaud's Phenomenon; Secondary Raynaud's Disease; Scleroderma; Raynaud's Disease secondary to systemic sclerosis; CREST; Apricus Biosciences; laser doppler; thermography
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Diffuse | interventions — Alprostadil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alprostadil Cream (300mcg) (Experimental): 300 micrograms/.42% Alprostadil Cream with 2.5% Dodecyl-2-N,N-dimethylaminopropionate hydrochloride (DDAIP-HCl) and Placebo, one dispenser for each administration
  Interventions: Drug: Alprostadil; Other: Placebo
- Alprostadil Cream (1000mcg) (Experimental): 1000 micrograms/.42% Alprostadil Cream with 2.5% Dodecyl-2-N,N-dimethylaminopropionate hydrochloride (DDAIP-HCl) and Placebo, one dispenser for each administration
  Interventions: Drug: Alprostadil; Other: Placebo
- Alprostadil Cream (3000mcg) (Experimental): 3000 micrograms/.42% Alprostadil Cream with 2.5% Dodecyl-2-N,N-dimethylaminopropionate hydrochloride (DDAIP-HCl) and Placebo, two dispensers for each administration
  Interventions: Drug: Alprostadil; Other: Placebo

INTERVENTIONS:
Drug: Alprostadil
Other: Placebo

SUMMARY:
The purpose of this study is to evaluate pharmacodynamics (PD) in adult subjects with a diagnosis of Raynaud's Phenomenon secondary to Systemic Sclerosis (SSc).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the pharmacodynamic (PD) effects of topical Alprostadil on digital perfusion by laser Doppler capillary velocimetry and digital temperature recovery with thermography following standardized cold challenge and to assess the safety and tolerability of 3 doses of Alprostadil topical cream and placebo cream in adult subjects with a diagnosis of Raynaud's Phenomenon secondary to Systemic Sclerosis (SSc).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of SSc by current ACR/EULAR Classification Criteria;
* Evidence of ongoing activity of Raynaud's Phenomenon as measured by a Raynaud Condition Score of 3 or greater at Screening;
* All females of childbearing potential must have a negative serum pregnancy test;

  a. Females of childbearing potential must abstain from sexual activity that could result in pregnancy, or agree to use an acceptable method of contraception throughout the study period and for 30 days following dosing of the investigational study drug. Acceptable contraception includes:
  1. Intrauterine devices
  2. Double barrier methods (e.g. condom or diaphragms with spermicidal gel or foam)
  3. Condom use is advised for all forms of contraception
* Must be willing and able to discontinue ongoing therapy for RP for at least 72 hours prior to each application of study medication; such drugs include calcium channel blockers, angiotensin-converting enzyme (ACE) inhibitors, short-acting PDE-5i (sildenafil, vardenafil, avanafil), sympatholytics and topical or systemic nitrates;
* Must be willing and able to discontinue consumption of caffeine-containing products (e.g., beverages and over-the-counter (OTC) medications) for at least 24 hours prior to each day of study dosing;
* Must be willing and able to remove jewelry from the treated hand prior to each day of study dosing;
* Must be willing to remove nail polish and/or nail coverings from the treated hand prior to each day of study dosing;
* Must not donate blood during the study;
* Have adequate finger extension to permit application of study treatments and attachment of physiologic measuring instruments.
* Must be willing to comply with all study procedures and study visits;
* Must provide written informed consent.

Exclusion Criteria:

* BMI less than 18.5;
* Clinically significant medical abnormality or history or presence of significant neurological, hepatic, renal, endocrine, gastrointestinal, cardiovascular, pulmonary, psychiatric and/or metabolic condition as determined by the Investigator);
* Clinical diagnosis of Systemic Sclerosis in association with other rheumatologic diseases including Mixed Connective Tissue Disease;
* Clinically significant abnormal laboratory test results at screening as determined by the Investigator;
* Raynaud's Phenomenon thought to be of non-systemic sclerosis etiology;
* Peripheral or central vasculopathy other than Systemic Sclerosis;
* History of Scleroderma renal crisis or currently being treated for hypertension, however, subjects with controlled hypertension will not be excluded;
* Active digital ulcers or rash on hand intended for study medication;
* History in the past (5) five years of autonomic neuropathy or postural hypotension;
* Upper extremity sympathectomy at any level in the 12 months prior to study;
* Tobacco smoking within six months of screening or unwillingness to avoid smoking throughout the study (e.g., cigarette, pipe, cigar, e-cigarettes) and the use of nicotine-containing products;
* Systolic Blood pressure less than 85mm/Hg;
* Prostanoid use by any route of administration within the previous six months;
* Current use of systemic or topical nitrates, endothelin receptor antagonists (e.g., bosentan) or any long-acting PDE-5 Inhibitors (e.g. tadalafil);
* Use of topical corticosteroid to the hand or fingers within 10 days of screening;
* Current use of ergot preparations, methysergide, B-adrenergic antagonists, contraceptives containing female steroid hormones, cyclosporine, clonidine, nicotine and cocaine;
* Pregnant or lactating female;
* Has known exaggerated pharmacological sensitivity or hypersensitivity to any drug similar to Alprostadil or its excipients;
* Has known hypersensitivity to nitrile;
* Involvement in any investigational drug or device study within 30 days prior to screening;
* History of non-compliance with treatment or clinic visit attendance.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic evaluation: digital perfusion by laser Doppler capillary velocimetry and on digital temperature recovery with thermography. | two hours (intermittently) after cold-challenge and post-dose
Safety assessments based on review of adverse events, vital sign measurements, electrocardiograms, physical examinations, and clinical laboratory tests. | One month

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Troupin, MD, MBA, Study Director — NEXMED (U.S.A.), Inc.
Locations (4):
- United States (4):
  - Diagnamics, Inc., Encinitas, California
  - University of Michigan Scleroderma Program - Division of Rheumatology/Dept. of Internal Medicine, Ann Arbor, Michigan
  - Cleveland Clinic, Cleveland, Ohio
  - Scleroderma Research Center - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania